CLINICAL TRIAL: NCT06918249
Title: Lupine Allergy in Children: Relevance of Sensitization and Severity of Reaction
Brief Title: Lupine Allergy in Children
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, ADAM Tania, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2025LAIC
Record Dates: First submitted 2025-03-30; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Food Allergy in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention

SUMMARY:
All children sensitized to lupine who have performed an oral food challenge (OFC) to lupine between January 2017 and May 2024 in the Pediatric Allergy Unit of the University Hospital of Nancy were included. Retrospective data regarding food and respiratory allergies were collected as well as information regarding lupine skin prick test (SPT), specific IgE (sIgE) and OFC. Severity of allergic reaction was evaluated by CoFAR grade and reactogenic cumulative threshold dose.

Aims of this study were (i) to assess relevance of sensitization to lupine in children and (ii) to describe severity of reactions in case of allergy.

ELIGIBILITY:
Inclusion Criteria:

* cutaneous or biological sensitization to lupine

Exclusion Criteria:

* oral food challenge done with something other than lupine flour

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children under 18 years as the study was done in the Pediatric Allergy department
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2024-05 (Actual); Study Completion 2024-05 (Actual)

PRIMARY OUTCOMES:
diagnostic value of prick test and specific IgE | baseline
  prick test to lupine flour in mm done during interview and collected retrospectively Specific IgE in kU/L to lupine seed done during same interview and collected retrospectively prick test and sIgE done as in usual clinical practice main outcome of the study are statistical tests (ROC curve) done to analyse diagnostic values of prick test and sIgE in this population

SECONDARY OUTCOMES:
severity of allergic reaction in oral food challenge | baseline
  grading the severity of allergic reaction in oral food challenge with lupine flour using CoFAR scale retrospectively

IPD SHARING:
Plan to Share IPD: Undecided